CLINICAL TRIAL: NCT02961881
Title: A Phase 1b Open-Label Study Investigating the Safety and Pharmacokinetics of Administration of Subcutaneous Blinatumomab for the Treatment of Relapsed/Refractory Indolent Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140286; 2016-002034-76 (EudraCT Number)
Record Dates: First submitted 2016-09-06; First posted 2016-11-11 (Estimated); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-05

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- blinatumomab (Experimental)
  Interventions: Drug: blinatumomab

INTERVENTIONS:
Drug: blinatumomab — Blinatumomab used as both continuous IV infusion and subcutaneous injection

SUMMARY:
Primary Objective:

• To evaluate the safety and tolerability of subcutaneous (SC) blinatumomab dose administrations

Secondary Objectives:

* To determine pharmacokinetics (PK) with continuous intravenous (cIV) and SC administrations
* To estimate the maximum tolerated dose (MTD) tested for blinatumomab administered subcutaneously
* To determine the incidence of anti-blinatumomab antibody formation following SC administration
* To evaluate efficacy response following treatment with SC blinatumomab administration

Exploratory Objective:

* To determine the pharmacodynamics (PD) time profiles for B-and T-lymphocytes as well as cytokine profiles during SC administration
* To evaluate efficacy response following treatment with SC blinatumomab administration using Lugano criteria if positron emission tomography-computed tomography (PET/CT) is used for evaluation

ELIGIBILITY:
Inclusion Criteria:

* Subject or subject's legally acceptable representative has provided informed consent.
* Age greater than or equal to 18 years old at the time of informed consent
* Subjects must have a histologically determined B cell NHL subtype as defined in the bullets below.

In addition, they must have disease that is primary refractory after initial therapy or have relapsed disease.

* Follicular Lymphoma I, II, IIIA
* Marginal zone lymphoma (extranodal, nodal or splenic). Subjects with gastric mucosa-
* associated lymphoid tissue must have progressed after Helicobacter pylori therapy and
* radiation. Subjects with splenic marginal zone lymphoma must have prior splenectomy.
* Lymphoplasmocytic lymphoma
* Mantle cell lymphoma ([MCL] with the exception of aggressive MCL, defined as Ki67 > 30%,
* or blastoid histology)
* Small lymphocytic lymphoma

  • Subjects without standard therapy alternatives, or contraindicated for standard therapy by investigator, or subjects unwilling to receive standard therapy. Disease status must be 1 of the following:
* Primary refractory (at least 1 prior line of therapy)
* Relapsed within 1 year of first response
* Responded to initial therapy for ≥ 1 year and relapsed after 2 or more lines of therapy, including an anti-CD20 monoclonal antibody

  * Measurable disease that has not been previously irradiated on positron emission tomography- computed tomography (PET-CT), or computed tomography (CT), of at least 1.5 cm within the last 21 days before the start of IP treatment.
  * Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
  * Life expectancy greater than or equal to 3 months as determined by treating physician.
  * Subjects must have adequate organ and marrow at screening as defined below:
* peripheral neutrophils >500/µL prior to start of treatment
* hemoglobin ≥8 g/dL
* Platelets greater than or equal to 50,000 mcL
* aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) < 5 × upper limit of normal (ULN
* Total bilirubin less than or equal to 1.5 x upper limit of normal (ULN)
* Creatinine clearance greater than or equal to 50 mL/min (Cockcroft-Gault)

Exclusion Criteria:

* Currently receiving treatment in another investigational device or drug study, or less than 30 days between ending treatment on another investigational device or drug study(ies) and start of IP treatment. Other investigational procedures while participating in this study are excluded.
* Known hypersensitivity to immunoglobulins or any other component of the study drug
* Subject likely to not be available to complete all protocol required study visits or procedures to the best of the subject and investigator's knowledge
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation procedures or completion.
* Subjects who have had treatments with anti-cancer agents including rituximab or obinutuzumab and/or other monoclonal antibody or radioimmunotherapy within 6 weeks before the starting IP treatment.
* Autologous stem cell transplantation within 12 weeks before the starting IP treatment or past history of allogeneic stem cell transplantation.
* Subjects who have received anti-CD 19 targeted therapies, chimeric antigen receptor T-cell or other cellular therapies for the treatment of their lymphoma .
* Subjects with suspected or known brain metastases should be excluded from this clinical study because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus or hepatitis C virus.
* History of or current relevant central nervous system pathology such as epilepsy, recurrent seizures, paresis, aphasia, apoplexia, severe brain injuries, cerebellar disease, organic brain syndrome or psychosis.
* History of malignancy other than their lymphoma with the exception of:

  * Malignancy treated with curative intent and with no known active disease present for ≥ 3 years before enrollment and felt to be at low risk for recurrence by the treating physician.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated cervical carcinoma in situ without evidence of disease.
  * Adequately treated breast ductal carcinoma in situ without evidence of disease
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer.
  * Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or uncontrolled systemic fungal bacteria, viral, or other infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* A female who is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 48 hours (Period 1) or 96 hours (Period 2), respectively, after the last dose of blinatumomab (Female subjects of childbearing potential should only be included in the study after a confirmed menstrual period and a negative highly sensitive urine or serum pregnancy test).
* A female of childbearing potential unwilling to use highly effective method of contraception during treatment and for an additional 48 hours (Period 1) or 96 hours (Period 2), respectively, after the last dose of blinatumomab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (17):
- United States (3):
  - City of Hope National Medical Center, Duarte, California
  - Rush University Medical Center, Chicago, Illinois
  - Hackensack University Medical Center, Hackensack, New Jersey
- Australia (3):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Epworth Healthcare, East Melbourne, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
- France (2):
  - Hopital Henri Mondor, CrÃ©teil Cedex
  - Hopital Saint Louis, Paris
- Germany (3):
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - UniversitÃ¤tsklinikum Frankfurt/Main, Frankfurt am Main
  - Universitatsklinikum Ulm, Ulm
- Italy (5):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Universitaria di Bologna Policlinico S Orsola Malpighi, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - IRCCS Ospedale San Raffaele, Milan
  - IRCCS Istituto Clinico Humanitas, Rozzano MI
- Leicester Royal Infirmary, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 39 participants screened, 35 participants were enrolled at 10 centers in the United States, Europe and Australia between 18 September 2017 and 02 September 2021.
Pre-assignment Details: The participants underwent an initial continuous intravenous (cIV) blinatumomab run-in period (Weeks 1 to 3). The participants received subcutaneous (SC) administration at Week 4 followed by a treatment free period of 2 to 3 days. After the SC administration period, participants received cIV treatment to complete 6 weeks of therapy (Weeks 5 to 6).
Groups:
- Blinatumomab Cohort 1: The participants underwent an initial cIV blinatumomab run-in period (Weeks 1 to 3) in which doses increased each week as follows: Week 1: 9 μq/day; Week 2: 28 μq/day; and Week 3: 112 μq/day. The run-in period was followed by a 12-hour treatment free period. The participants then received 112 μq SC administrations every 12 hours (q12h) for 5 days at Week 4 followed by a treatment free period of 2 to 3 days. After the SC administration period, the participants received 112 μq/day cIV blinatumomab during Weeks 5 and 6.
- Blinatumomab Cohort 2: The participants underwent an initial cIV blinatumomab run-in period (Weeks 1 to 3) in which doses increased each week as follows: Week 1: 9 μq/day; Week 2: 28 μq/day; and Week 3: 112 μq/day. The run-in period was followed by a 12-hour treatment free period. The participants then received 225 μq SC administrations q12h for 5 days at Week 4 followed by a treatment free period of 2 to 3 days. After the SC administration period, the participants received 112 μq/day cIV blinatumomab during Weeks 5 and 6.
- Blinatumomab Cohort 3: The participants underwent an initial cIV blinatumomab run-in period (Weeks 1 to 3) in which doses increased each week as follows: Week 1: 9 μq/day; Week 2: 28 μq/day; and Week 3: 112 μq/day. The run-in period was followed by a 12-hour treatment free period. The participants then received 450 μq SC administrations every 24 hours (q24h) for 5 days at Week 4 followed by a treatment free period of 2 to 3 days. After the SC administration period, the participants received 112 μq/day cIV blinatumomab during Weeks 5 and 6.
- Blinatumomab Cohort 4: The participants underwent an initial cIV blinatumomab run-in period (Weeks 1 to 3) in which doses increased each week as follows: Week 1: 9 μq/day; Week 2: 28 μq/day; and Week 3: 112 μq/day. The run-in period was followed by a 12-hour treatment free period. The participants then received 675 μq SC administrations q24h for 5 days at Week 4 followed by a treatment free period of 2 to 3 days. After the SC administration period, the participants received 112 μq/day cIV blinatumomab during Weeks 5 and 6.
- Blinatumomab Cohort 5: The participants underwent an initial cIV blinatumomab run-in period (Weeks 1 to 3) in which doses increased each week as follows: Week 1: 9 μq/day; Week 2: 28 μq/day; and Week 3: 112 μq/day. The run-in period was followed by a 12-hour treatment free period. The participants then received 675 μq SC administrations every 48 hours (q48h) for 5 days at Week 4 followed by a treatment free period of 2 to 3 days. After the SC administration period, the participants received 112 μq/day cIV blinatumomab during Weeks 5 and 6.
Period: Overall Study
Arm/Group | Blinatumomab Cohort 1 | Blinatumomab Cohort 2 | Blinatumomab Cohort 3 | Blinatumomab Cohort 4 | Blinatumomab Cohort 5
Started | 7 | 8 | 8 | 6 | 6
Started Week 4 SC Dosing | 6 | 7 | 7 | 6 | 5
Started Week 5-6 cIV Dosing | 6 | 5 | 6 | 6 | 5
Completed (Participants who completed investigational product) | 5 | 4 | 5 | 6 | 5
Not Completed | 2 | 4 | 3 | 0 | 1
Not completed — Adverse Event | 1 | 2 | 2 | 0 | 1
Not completed — Participant request | 0 | 2 | 0 | 0 | 0
Not completed — Disease progression | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Blinatumomab Cohort 1: The participants underwent an initial cIV blinatumomab run-in period (Weeks 1 to 3) in which doses increased each week as follows: Week 1: 9 μq/day; Week 2: 28 μq/day; and Week 3: 112 μq/day. The run-in period was followed by a 12-hour treatment free period. The participants then received 112 μq SC administrations q12h for 5 days at Week 4 followed by a treatment free period of 2 to 3 days. After the SC administration period, the participants received 112 μq/day cIV blinatumomab during Weeks 5 and 6.
- Blinatumomab Cohort 3: Blinatumomab Cohort 3 The participants underwent an initial cIV blinatumomab run-in period (Weeks 1 to 3) in which doses increased each week as follows: Week 1: 9 μq/day; Week 2: 28 μq/day; and Week 3: 112 μq/day. The run-in period was followed by a 12-hour treatment free period. The participants then received 450 μq SC administrations q24h for 5 days at Week 4 followed by a treatment free period of 2 to 3 days. After the SC administration period, the participants received 112 μq/day cIV blinatumomab during Weeks 5 and 6.
- Blinatumomab Cohort 5: The participants underwent an initial cIV blinatumomab run-in period (Weeks 1 to 3) in which doses increased each week as follows: Week 1: 9 μq/day; Week 2: 28 μq/day; and Week 3: 112 μq/day. The run-in period was followed by a 12-hour treatment free period. The participants then received 675 μq SC administrations q48h for 5 days at Week 4 followed by a treatment free period of 2 to 3 days. After the SC administration period, the participants received 112 μq/day cIV blinatumomab during Weeks 5 and 6.
- Total: Total of all reporting groups
Arm/Group | Blinatumomab Cohort 1 | Blinatumomab Cohort 2 | Blinatumomab Cohort 3 | Blinatumomab Cohort 4 | Blinatumomab Cohort 5 | Total
Number analyzed (Participants) | 7 | 8 | 8 | 6 | 6 | 35
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 5 | 5 | 3 | 3 | 5 | 21
  65 - 74 years | 2 | 2 | 5 | 3 | 1 | 13
  75 - 84 years | 0 | 1 | 0 | 0 | 0 | 1
  ≥ 85 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 3 | 1 | 16
  Male | 4 | 4 | 3 | 3 | 5 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 6 | 7 | 8 | 6 | 6 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Black (or African American) | 1 | 0 | 0 | 0 | 0 | 1
  Multiple | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 7 | 8 | 6 | 6 | 31
  Other | 2 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting-Toxicities (DLTs) After SC Administration
Description: The occurrence of any of the following toxicities during the DLT evaluation period was considered a DLT, if judged by the investigator to be related to the administration of blinatumomab:
  * Death
  * Any toxicity, regardless of grade, that lead to a participant's removal from the study by the investigator and/or sponsor
  * Persistent Common Terminology Criteria for Adverse Events (CTCAE) grade >/= 2 non-hematologic adverse events (AEs) that were deemed intolerable by the participant or the treating physician and that did not respond to appropriate medical management within 5 days and lead to treatment discontinuation
  * Recurrent grade 2 seizures
  * All grade 3 and 4 AEs and laboratory abnormalities, which occurred during the SC administration portion of the treatment period with exceptions noted in protocol section 6.2.1.2.3.
Time Frame: Day 1 to Day 7 of Week 4
Population: DLT analysis set included DLT-evaluable participants who received all (q48h dosing), >/= 4/5 (q24h dosing) or >/= 8/9 (q12h dosing) doses of SC blinatumomab or experienced a DLT during the DLT evaluable period.
Measure: Count of Participants; unit: Participants
Groups:
- Blinatumomab SC Cohort 1: The participants received 112 μq SC administrations q12h for 5 days at Week 4 followed by a treatment free period of 2 to 3 days.
- Blinatumomab SC Cohort 2: The participants received 225 μq SC administrations q12h for 5 days at Week 4 followed by a treatment free period of 2 to 3 days.
- Blinatumomab SC Cohort 3: The participants received 450 μq SC administrations q24h for 5 days at Week 4 followed by a treatment free period of 2 to 3 days.
- Blinatumomab SC Cohort 4: The participants received 675 μq SC administrations q24h for 5 days at Week 4 followed by a treatment free period of 2 to 3 days.
- Blinatumomab SC Cohort 5: The participants received 675 μq SC administrations q48h for 5 days at Week 4 followed by a treatment free period of 2 to 3 days.
Arm/Group | Blinatumomab SC Cohort 1 | Blinatumomab SC Cohort 2 | Blinatumomab SC Cohort 3 | Blinatumomab SC Cohort 4 | Blinatumomab SC Cohort 5
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 5
Participants | 0 | 1 | 1 | 0 | 0

2. Primary Outcome: Number of Participants With DLTs CTCAE Grade ≥ 3 After SC Administration
Description: All toxicities were graded using the CTCAE version 4.0: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = fatal.
Time Frame: Day 1 to Day 7 of Week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab SC Cohort 1 | Blinatumomab SC Cohort 2 | Blinatumomab SC Cohort 3 | Blinatumomab SC Cohort 4 | Blinatumomab SC Cohort 5
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 5
Participants | 0 | 1 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) After SC Administration
Description: An AE was defined as any untoward medical occurrence in a clinical study participant. The AE did not necessarily have a causal relationship with study treatment. The definition of AEs included worsening of a pre-existing medical condition.
  TEAEs included AEs starting on or after first dose of investigational product and up to the end of study date. All AEs were graded using the CTCAE version 4.0: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = fatal.
Time Frame: Day 1 to end of study (approximately 17 weeks)
Population: Safety analysis set included participants that were enrolled and received at least 1 dose of blinatumomab.
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab SC Cohort 1 | Blinatumomab SC Cohort 2 | Blinatumomab SC Cohort 3 | Blinatumomab SC Cohort 4 | Blinatumomab SC Cohort 5
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 5
Participants
  Any TEAEs | 2 | 6 | 6 | 6 | 4
  Any TEAEs CTCAE Grade ≥ 3 | 1 | 1 | 2 | 1 | 0

4. Secondary Outcome: Steady State Serum Concentration (Css) of Blinatumomab After cIV Administration
Description: Summarized as the observed concentrations collected after 5 half-lives after the start of the IV infusion of each dose (i.e., 9, 28 and 112 μg/day).
Time Frame: Once at any timepoint during Day 2 of Weeks 1, 2, 3, 5 and 6
Population: Pharmacokinetic (PK) analyses set included all participants who received any cIV blinatumomab and had at least one PK sample. These participants were evaluated for PK unless significant protocol deviations affected the data analysis or if key dosing, dosing interruption, or sampling information was missing. Css data during cIV dosing was reported per dose level as pre-specified in statistical analysis plan (SAP) section 10.7.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Groups:
- Blinatumomab cIV Before SC Week 1: The participants received 9 μq/day cIV administrations during Week 1.
- Blinatumomab cIV Before SC Week 2: The participants received 28 μq/day cIV administrations during Week 2.
- Blinatumomab cIV Before SC Week 3: The participants received 112 μq/day cIV administrations during Week 3.
- Blinatumomab cIV After SC: After the SC administration period, the participants received 112 μq/day cIV blinatumomab during Weeks 5 and 6.
Arm/Group | Blinatumomab cIV Before SC Week 1 | Blinatumomab cIV Before SC Week 2 | Blinatumomab cIV Before SC Week 3 | Blinatumomab cIV After SC
Number analyzed (Participants) | 29 | 31 | 29 | 26
pg/mL | 238 (137) | 672 (94) | 2780 (87) | 2700 (85)

5. Secondary Outcome: Systemic Clearance (CL) of Blinatumomab After cIV Administration
Description: Calculated as CL=R0/Css; where R0 is the infusion rate (μg/hr) and Css is the average Css. Both R0 and Css were dose-normalized to 112 μg/day for this calculation.
Time Frame: Once at any timepoint during Day 2 of Weeks 1, 2, 3, 5 and 6
Population: PK analyses set included all participants who received any cIV blinatumomab and had at least one PK sample. These participants were evaluated for PK unless significant protocol deviations affected the data analysis or if key dosing, dosing interruption, or sampling information was missing. CL data prior to SC dosing was dose-normalized and reported together as pre-specified in SAP section 10.7.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Groups:
- Blinatumomab cIV Before SC: The participants underwent an initial cIV blinatumomab run-in period (Weeks 1 to 3) in which doses increased each week as follows: Week 1: 9 μq/day; Week 2: 28 μq/day; and Week 3: 112 μq/day.
Arm/Group | Blinatumomab cIV Before SC | Blinatumomab cIV After SC
Number analyzed (Participants) | 33 | 26
L/hr | 1.67 (111) | 1.73 (85)

6. Secondary Outcome: Maximum Observed Concentration (Cmax) of Blinatumomab After SC Administration
Time Frame: Week 4 Day 1 (pre-dose and 1, 2, 4, 6, 8 and 12 hours post-dose) and Week 4 Day 5 (pre-dose and 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose)
Population: PK analyses set included all participants who received any SC blinatumomab and had at least one PK sample. These participants were evaluated for PK unless significant protocol deviations affected the data analysis or if key dosing, dosing interruption, or sampling information was missing. Descriptive statistics for first SC dose of 675 μg on Week 4 Day 1 were determined using parameter estimates from participants in Cohorts 4 and 5 as pre-specified in SAP section 10.7.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Groups:
- Blinatumomab SC Cohorts 4 and 5: The participants received 675 μq SC administrations q24h or q48h for 5 days at Week 4 followed by a treatment free period of 2 to 3 days.
Arm/Group | Blinatumomab SC Cohort 1 | Blinatumomab SC Cohort 2 | Blinatumomab SC Cohort 3 | Blinatumomab SC Cohorts 4 and 5 | Blinatumomab SC Cohort 4 | Blinatumomab SC Cohort 5
Number analyzed (Participants) | 6 | 7 | 7 | 10 | 6 | 4
pg/mL
  Week 4 Day 1: number analyzed (Participants) | 6 | 7 | 7 | 10 | 0 | 0
  Week 4 Day 1 | 877 (88) | 1810 (93) | 2650 (98) | 4260 (103) |  |
  Week 4 Day 5: number analyzed (Participants) | 6 | 5 | 6 | 0 | 6 | 4
  Week 4 Day 5 | 2070 (15) | 4340 (36) | 4290 (98) |  | 5690 (71) | 4340 (304)

7. Secondary Outcome: Time at Which Cmax (Tmax) Occurred of Blinatumomab After SC Administration
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Blinatumomab SC Cohort 1 | Blinatumomab SC Cohort 2 | Blinatumomab SC Cohort 3 | Blinatumomab SC Cohorts 4 and 5 | Blinatumomab SC Cohort 4 | Blinatumomab SC Cohort 5
Number analyzed (Participants) | 6 | 7 | 7 | 10 | 6 | 4
hours
  Week 4 Day 1: number analyzed (Participants) | 6 | 7 | 7 | 10 | 0 | 0
  Week 4 Day 1 | 5.0 [0.0 to 8.1] | 7.9 [1.0 to 8.1] | 12 [7.2 to 12] | 12 [1.9 to 12] |  |
  Week 4 Day 5: number analyzed (Participants) | 6 | 5 | 6 | 0 | 6 | 4
  Week 4 Day 5 | 2.8 [0.0 to 8.0] | 4.0 [0.0 to 6.1] | 7.6 [6.0 to 12] |  | 8.0 [4.0 to 12] | 9.5 [2.2 to 12]

8. Secondary Outcome: Area Under the Concentration-time Curve (AUC) of Blinatumomab After SC Administration for a Dosing Interval t (AUCt)
Description: Estimated using the linear trapezoidal method; where t is a dosing interval. AUC over the dosing interval, t where t is 12 hours for Cohorts 1 and 2, 24 hours for Cohorts 3 and 4, and 48 hours for Cohort 5.
Time Frame: as for outcome 6
Population: PK analyses set included all participants who received any SC blinatumomab and had at least one PK sample. These participants were evaluated for PK unless significant protocol deviations affected the data analysis or if key dosing, dosing interruption, or sampling information was missing. At Week 4 Day 1, AUCt was only reported for SC dosing regimens in Cohorts 1 and 2 as PK sampling was taken only over the 12-hour period following dosing as pre-specified in protocol section 7.1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr•pg/mL
Arm/Group | Blinatumomab SC Cohort 1 | Blinatumomab SC Cohort 2 | Blinatumomab SC Cohort 3 | Blinatumomab SC Cohort 4 | Blinatumomab SC Cohort 5
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 4
hr•pg/mL
  Week 4 Day 1: number analyzed (Participants) | 5 | 2 | 0 | 0 | 0
  Week 4 Day 1 | 6080 (80) | 9430 (40) |  |  |
  Week 4 Day 5 | 19100 (21) | 40500 (41) | 72000 (92) | 90900 (77) | 90800 (236)

9. Secondary Outcome: Minimum Observed Concentration (Cmin) of Blinatumomab After SC Administration
Time Frame: as for outcome 6
Population: PK analyses set included all participants who received any SC blinatumomab and had at least one PK sample. These participants were evaluated for PK unless significant protocol deviations affected the data analysis or if key dosing, dosing interruption, or sampling information was missing. At Week 4 Day 1, Cmin was only reported for SC dosing regimens in Cohorts 1 and 2 as PK sampling was taken only over the 12-hour period following dosing as pre-specified in protocol section 7.1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Blinatumomab SC Cohort 1 | Blinatumomab SC Cohort 2 | Blinatumomab SC Cohort 3 | Blinatumomab SC Cohort 4 | Blinatumomab SC Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4
pg/mL
  Week 4 Day 1: number analyzed (Participants) | 6 | 6 | 0 | 0 | 0
  Week 4 Day 1 | 651 (93) | 1470 (101) |  |  |
  Week 4 Day 5: number analyzed (Participants) | 6 | 5 | 6 | 6 | 4
  Week 4 Day 5 | 1290 (30) | 2550 (41) | 1950 (94) | 2130 (104) | 147 (66)

10. Secondary Outcome: Apparent Clearance (CL/F) of Blinatumomab After SC Administration
Description: Calculated as CL/F = Dose sc / AUCt-ss (at steady state).
Time Frame: Week 4 Day 5 (pre-dose and 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose)
Population: PK analyses set included all participants who received any SC blinatumomab and had at least one PK sample. These participants were evaluated for PK unless significant protocol deviations affected the data analysis or if key dosing, dosing interruption, or sampling information was missing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Blinatumomab SC Cohort 1 | Blinatumomab SC Cohort 2 | Blinatumomab SC Cohort 3 | Blinatumomab SC Cohort 4 | Blinatumomab SC Cohort 5
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 4
L/hr | 5.85 (21) | 5.55 (41) | 6.25 (92) | 7.43 (77) | 7.43 (236)

11. Secondary Outcome: Volume of Distribution Based on Terminal Phase (Vz/F) of Blinatumomab After SC Administration
Description: Calculated as Vz/F=CL/F / λz, where λz was the first-order rate constant estimated via linear regression of the terminal log-linear decay phase as determined from the noncompartmental analysis.
Time Frame: Week 4 Day 5 (pre-dose and 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Blinatumomab SC Cohort 1 | Blinatumomab SC Cohort 2 | Blinatumomab SC Cohort 3 | Blinatumomab SC Cohort 4 | Blinatumomab SC Cohort 5
Number analyzed (Participants) | 6 | 5 | 3 | 4 | 2
liters | 83.4 (19) | 100 (93) | 58.6 (115) | 120 (97) | 133 (9623)

12. Secondary Outcome: Terminal Half-life (t1/2,z) of Blinatumomab After SC Administration
Description: Calculated as t1/2,z = ln(2) / λz.
Time Frame: Week 4 Day 5 (pre-dose and 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Blinatumomab SC Cohort 1 | Blinatumomab SC Cohort 2 | Blinatumomab SC Cohort 3 | Blinatumomab SC Cohort 4 | Blinatumomab SC Cohort 5
Number analyzed (Participants) | 6 | 4 | 3 | 4 | 2
hours | 9.87 (12) | 10.7 (22) | 7.30 (21) | 11.7 (30) | 9.20 (83)

13. Secondary Outcome: Accumulation Ratio of Blinatumomab After SC Administration
Description: Calculated as the ratio of AUCt (last SC dose; Week 4 Day 5) / AUC (first SC dose; Week 4 Day 1).
Time Frame: as for outcome 6
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Blinatumomab SC Cohort 1 | Blinatumomab SC Cohort 2 | Blinatumomab SC Cohort 3 | Blinatumomab SC Cohort 4 | Blinatumomab SC Cohort 5
Number analyzed (Participants) | 5 | 2 | 2 | 5 | 3
ratio | 3.25 (61) | 4.14 (35) | 2.31 (63) | 1.71 (109) | 1.01 (107)

14. Secondary Outcome: Bioavailability (F) of SC Blinatumomab
Description: Calculated as F = (CL * AUCt-ss) / Dose sc.
Time Frame: Week 4 Day 5 (pre-dose and 1, 2, 4, 6, 8, 12, 24 and 48 hours post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent bioavailability
Arm/Group | Blinatumomab SC Cohort 1 | Blinatumomab SC Cohort 2 | Blinatumomab SC Cohort 3 | Blinatumomab SC Cohort 4 | Blinatumomab SC Cohort 5
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 4
percent bioavailability | 32.1 (38) | 22.5 (54) | 33.8 (215) | 24.6 (53) | 30.2 (180)

15. Secondary Outcome: Maximum Tolerated Dose (MTD) of SC Blinatumomab
Description: The MTD was defined as the highest dose level at which </= 1 of 6 participants experienced a DLT.
Time Frame: Day 1 to Day 7 of Week 4
Population: DLT analysis set included all DLT-evaluable participants who received all doses (q48h), at least 4/5 doses (q24h) or at least 8/9 doses (q12h) of SC blinatumomab.
Measure: Number; unit: μq
Groups:
- Blinatumomab SC Total: The participants received SC administrations for 5 days at Week 4 followed by a treatment free period of 2 to 3 days.
Arm/Group | Blinatumomab SC Total
Number analyzed (Participants) | 30
μq | NA — The MTD was not reached in this study.

16. Secondary Outcome: Number of Participants With Anti-blinatumomab Antibody Formation After SC Administration
Time Frame: Predose at the re-start of cIV infusion (Week 5 Day 1)
Population: Safety analysis set included participants that were enrolled and received at least 1 dose of blinatumomab.
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab SC Cohort 1 | Blinatumomab SC Cohort 2 | Blinatumomab SC Cohort 3 | Blinatumomab SC Cohort 4 | Blinatumomab SC Cohort 5
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 5
Participants | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Overall Response Rate (ORR) After SC Administration
Description: Percentage of participants achieving ORR (complete response [CR] + partial response [PR]) was determined by best overall response using Cheson criteria:
  * CR: disappearance of all evidence of disease.
  * PR: regression of measurable disease and no new sites.
  The 95% confidence interval (CI) was calculated using Clopper-Pearson exact CI. Participants were considered as non-responders if there was no response assessment available.
Time Frame: Day 1 to end of study (approximately 17 weeks)
Population: Full analysis set included participants that were enrolled and received at least 1 dose of blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab SC Cohort 1 | Blinatumomab SC Cohort 2 | Blinatumomab SC Cohort 3 | Blinatumomab SC Cohort 4 | Blinatumomab SC Cohort 5
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 5
percentage of participants | 66.7 [22.3 to 95.7] | 71.4 [29.0 to 96.3] | 71.4 [29.0 to 96.3] | 83.3 [35.9 to 99.6] | 40.0 [5.3 to 85.3]

ADVERSE EVENTS:
Time Frame: Day 1 to end of study (approximately 17 weeks)
Description: Safety analysis set included participants that were enrolled and received at least 1 dose of blinatumomab.
Groups:
- Blinatumomab cIV Total: The participants underwent an initial cIV blinatumomab run-in period (Weeks 1 to 3) in which doses increased each week as follows: Week 1: 9 μq/day; Week 2: 28 μq/day; and Week 3: 112 μq/day. After the SC administration period, the participants received 112 μq/day cIV blinatumomab during Weeks 5 and 6.
- Blinatumomab SC + cIV Total: The participants underwent an initial cIV blinatumomab run-in period (Weeks 1 to 3) in which doses increased each week as follows: Week 1: 9 μq/day; Week 2: 28 μq/day; and Week 3: 112 μq/day. The run-in period was followed by a 12-hour treatment free period. The participants then received SC administrations for 5 days at Week 4 followed by a treatment free period of 2 to 3 days. After the SC administration period, the participants received 112 μq/day cIV blinatumomab during Weeks 5 and 6.
Arm/Group | Blinatumomab cIV Before SC Week 1 | Blinatumomab cIV Before SC Week 2 | Blinatumomab cIV Before SC Week 3 | Blinatumomab SC Cohort 1 | Blinatumomab SC Cohort 2 | Blinatumomab SC Cohort 3 | Blinatumomab SC Cohort 4 | Blinatumomab SC Cohort 5 | Blinatumomab cIV After SC | Blinatumomab SC Total | Blinatumomab cIV Total | Blinatumomab SC + cIV Total
All-Cause Mortality (participants affected / at risk) | 1/35 | 0/34 | 0/33 | 0/6 | 0/7 | 0/7 | 0/6 | 0/5 | 1/28 | 0/31 | 2/35 | 2/35
Serious Adverse Events (participants affected / at risk) | 5/35 | 5/34 | 8/33 | 0/6 | 1/7 | 1/7 | 0/6 | 0/5 | 10/28 | 2/31 | 18/35 | 19/35
Other Adverse Events (participants affected / at risk) | 23/35 | 22/34 | 23/33 | 2/6 | 6/7 | 6/7 | 6/6 | 4/5 | 19/28 | 24/31 | 34/35 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab cIV Before SC Week 1 (N=35) | Blinatumomab cIV Before SC Week 2 (N=34) | Blinatumomab cIV Before SC Week 3 (N=33) | Blinatumomab SC Cohort 1 (N=6) | Blinatumomab SC Cohort 2 (N=7) | Blinatumomab SC Cohort 3 (N=7) | Blinatumomab SC Cohort 4 (N=6) | Blinatumomab SC Cohort 5 (N=5) | Blinatumomab cIV After SC (N=28) | Blinatumomab SC Total (N=31) | Blinatumomab cIV Total (N=35) | Blinatumomab SC + cIV Total (N=35)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Dermo-hypodermitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Device related sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Marginal zone lymphoma refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Coordination abnormal (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Motor dysfunction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 4
Neurological symptom (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neurotoxicity (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab cIV Before SC Week 1 (N=35) | Blinatumomab cIV Before SC Week 2 (N=34) | Blinatumomab cIV Before SC Week 3 (N=33) | Blinatumomab SC Cohort 1 (N=6) | Blinatumomab SC Cohort 2 (N=7) | Blinatumomab SC Cohort 3 (N=7) | Blinatumomab SC Cohort 4 (N=6) | Blinatumomab SC Cohort 5 (N=5) | Blinatumomab cIV After SC (N=28) | Blinatumomab SC Total (N=31) | Blinatumomab cIV Total (N=35) | Blinatumomab SC + cIV Total (N=35)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 5 | 6
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 6 | 1 | 8 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 4 | 5
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 3 | 3
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 6 | 3 | 4 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 13 | 14
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 5 | 1 | 8 | 8
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 5 | 6
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 3
Administration site erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Asthenia (General disorders) | 2 | 4 | 2 | 0 | 0 | 1 | 1 | 0 | 5 | 2 | 7 | 7
Fatigue (General disorders) | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 5 | 5
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 4 | 4
Pyrexia (General disorders) | 7 | 3 | 11 | 1 | 0 | 1 | 0 | 0 | 4 | 2 | 17 | 18
Cytokine release syndrome (Immune system disorders) | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 4 | 4 | 6
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Oral herpes (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 4
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 3
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 3
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 4 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 4 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 5 | 5
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 2 | 3
Cognitive disorder (Nervous system disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 2 | 2
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Dysgraphia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 3
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Headache (Nervous system disorders) | 4 | 3 | 6 | 0 | 2 | 1 | 0 | 0 | 7 | 3 | 15 | 16
Nervous system disorder (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 4
Neurotoxicity (Nervous system disorders) | 3 | 1 | 3 | 1 | 1 | 0 | 2 | 0 | 2 | 4 | 5 | 7
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 2
Subdural hygroma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 4 | 1 | 9 | 0 | 0 | 0 | 2 | 0 | 4 | 2 | 12 | 12
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Confusional state (Psychiatric disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Insomnia (Psychiatric disorders) | 3 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 3 | 7 | 9
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 3
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Astringent therapy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT02961881/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT02961881/SAP_001.pdf